CLINICAL TRIAL: NCT07089342
Title: Exploring Biological Markers of Driver Fatigue for Enhanced Road Safety
Acronym: FATIGUE
Status: Recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Vias Institute Brussel (Unknown); Nationaal Instituut voor Criminalistiek en Criminologie Brussel (Unknown)
Responsible Party: Sponsor
Other Study IDs: EC-2025-141; EC-2025-141 (Other: COMMISSIE MEDISCHE ETHIEK BRUSSEL)
Record Dates: First submitted 2025-07-09; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Drowsiness; Sleepiness; Fatigue
Keywords: Fatigue; Drowsy driving; Sleepiness; Road Safety
MeSH Terms: conditions — Sleepiness; Fatigue

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — oral fluid/saliva
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Road traffic population: People randomly stopped by police in public road traffic

SUMMARY:
The aim of this study is to assess the effectiveness of biological markers in detecting fatigue/sleepiness in a sample of the general driving population in Belgium. The link between the collected biomarkers (oral fluid sample), observed signs of sleepiness in the driver and self-reported driver variables will be analysed. The analysis of the biological samples aims to measure endogenous metabolite levels that are possibly indicative for sleepiness of the donor driver. The respective metabolites will be chosen based on the results of a preceding clinical study (https://clinicaltrials.gov/study/NCT05585515). The objective of this study is to verify and validate the proposed metabolites as biomarkers for driver sleepiness in road traffic.

DETAILED DESCRIPTION:
Researchers from NICC (National Institute of Criminalistics and Criminology) and VIAS will collect (1) saliva samples (Salivette with neutral swab allowing use by not-medically trained personnel; this sampling method is also used by the Belgian police in scope of the drugs in traffic legislation since 2019), (2) self-reported driver data (survey) and (3) observed driver data (form filled in by researchers) from drivers that were stopped on the road in scope of routine police checks. The collaboration with the police is because police can stop drivers randomly on-road while researchers cannot. After the police check, a researcher will ask if the driver wants to participate in a study on driver fatigue which is entirely independent from the police check. Voluntary drivers sign an informed consent form.

The collected saliva samples will be entirely separate from any sample obtained during the police checks. During data collection, the saliva sample, driver survey and observation form will each get a unique identification code to link the data. Afterwards, the researchers will work with this anonymised number and the data cannot be traced back to the participant.

All anonymised samples/data will temporarily be stored at NICC (Dept. Toxicology) and then be sent to the University of Zurich for analysis. The analysis of the saliva samples aims to measure endogenous metabolite levels that are possibly indicative for sleepiness of the donor. The correlation of the biomarker levels with observed/reported driver data will be measured. In specific cases the co-existence of drugs/medication in the saliva samples may also be tested: when the donor reported the consumption of the respective substance in the driver survey, as a confirmatory analysis, and (2) when the researchers believe the co-consumption of drugs/medication may interfere with the primary analysis. All anonymised samples will be stored at the University of Zurich for a maximum of 10 years and then be destroyed.

ELIGIBILITY:
Inclusion Criteria:

* drivers randomly stopped by the police

Exclusion Criteria:

* refusal to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Drivers (all vehicle types, aged 18 or older) voluntarily participating after being randomly stopped during roadside police checks in Belgium
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes in metabolite concentrations in oral fluid quantified by liquid chromatography with mass spectrometry | Baseline: One collection time point after enrollment
  Investigators will collect oral fluid samples for quantification of all detectable metabolites. Investigators will analyze which metabolite concentration values undergo significant changes with regard to sleep/wake history and demographical data of the donor.

SECONDARY OUTCOMES:
Subjective sleepiness | Baseline: One time point after enrollment
  Participants will complete the Karolinska Sleepiness Scale (version A) questionnaire. It is a 9-point scale, ranging from 1 (extremely alert) to 9 (very sleepy, great effort to keep awake, fighting sleep).
Behavioral markers of drowsy driving: Shivering | Baseline: One time point after enrollment
  Investigators will examine participants for behavioral abnormalities concerning shivering based on this scale: (i) yes (ii) no (iii) uncertain
Behavioral markers of drowsy driving: Reaction | Baseline: One time point after enrollment
  Investigators will examine participants for behavioral abnormalities concerning reaction based on this scale: (i) slow/tired (ii) normal (iii) fast/talkative
Behavioral markers of drowsy driving: Gait | Baseline: One time point after enrollment
  Investigators will examine participants for behavioral abnormalities concerning gait based on this scale: (i) slow (ii) normal (iii) uncertain

CONTACTS AND LOCATIONS:
Locations (1):
- Vias institute, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
Results will be published in peer-reviewed journals. Anonymized raw data will be made available upon request.